CLINICAL TRIAL: NCT07091721
Title: The Mentalization Intervention for Children and Adolescents (MICA) Study: A Randomised Controlled Trial of Support for Aggressive and Violent Behaviour Via Forensic Child and Adolescent Mental Health Services (FCAMHS)
Brief Title: Using Mentalization Based Therapy to Support Children and Adolescents Referred to Specialist Mental Health Services in the NHS for Aggressive and/or Violent Behaviour
Acronym: MICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Freud (Other)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Julian Edbrooke-Childs, Co-Director of Evidence Based Practice Unit, Anna Freud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBTCD01
Record Dates: First submitted 2025-07-14; First posted 2025-07-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-07

CONDITIONS: Conduct Disorder; Mentalization Based Therapy; Violent Behavior; Aggressive Behaviour; Adolescent Behavior; Children Behavior
Keywords: The Mentalization Intervention for Children and Adolescents (MICA) study.; Forensic Child and Adolescent Mental Health Services (FCAMHS).; Aggressive and violent behaviour.; Mentalization-Based Therapy.; Conduct disorder.; Mental Health.; Young people.; MBT-CD
MeSH Terms: conditions — Conduct Disorder; Aggression; Adolescent Behavior; Psychological Well-Being | interventions — Mentalization-Based Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBT (Experimental)
  Interventions: Behavioral: Mentalization based therapy (MBT)
- Support as usual (Active Comparator)
  Interventions: Other: Support as usual

INTERVENTIONS:
Behavioral: Mentalization based therapy (MBT) — Mentalization based therapy for conduct disorder
  Arms: MBT
Other: Support as usual — Support usually provided by FCAMHS which may include advice/guidance to the professional network around the child/adolescent, psychoeducation, other mental health treatment e.g. CBT
  Arms: Support as usual

SUMMARY:
The MICA Study is a research project that has been designed to work out how helpful mentalisation based therapy is. This is a new type of support that helps young people make sense of their own behaviours and feelings, and those of others. It involves meeting regularly with a mental health practitioner and parents/carers can be involved in some meetings too. It is hoped that this new type of support will help young people stop acting aggressively/violently.

This project will be delivered in Forensic Child and Adolescent Mental Health Services (FCAMHS) in England. This service supports some of the most vulnerable young people in the country, who may also have involvement from other professionals including the Youth Justice System.

The aim of the research is to make the support better for young people who use these services. This research involves doing a randomised controlled trial. This means half the young people will get the usual support from FCAMHS, and half will get the usual support plus the new support. The results will be used to compare mentalisation based therapy to the support FCAMHS usually provides. This will show the best way to support young people with their aggressive/violent behaviours.

To start with, young people will answer a questionnaire. Following this, young people will receive either usual support or usual support plus MBT for six months. After this, young people will answer a questionnaire again. Some young people will be asked to take part in an optional interview to share their thoughts on this research. All young people aged 10-17 years who have been referred to a FCAMHS in England will be asked to take part, as long as they can speak and understand English. Some young people might not want to take part in this research and that will not change the support they receive.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 years at the time of referral;
* Aggression and/or violence are indicated at referral or assessment;
* Participation in the evaluation would not interfere with statutory orders;
* Child and parent/carer (for children 10-15 years) are able to consent and engage with the study materials;
* Living in the community at time of referral and no imminent plans to move to hospital, residential, or secure settings.

Additional inclusion criteria for participants recruited from a clinician's existing caseload:

* There has been no direct contact between child and FCAMHS clinicians, including assessments.
* There has been no indirect therapeutic support provided by FCAMHS e.g. advising non-FCAMHS professionals on therapeutic support.
* It is permissible for the clinician to have previously engaged in consultation activities where these did not involve contact with the child.

Exclusion Criteria:

* Age under 10 or age 18 or older at the time of referral;
* No evidence of aggression and/or violence indicated at referral or assessment;
* FCAMHS are only offering a one-off consultation or assessment (e.g., the network around the child requires support to manage risk but additional input is not required);
* Child's level of English is not sufficient to engage in the intervention;
* Child and/or parents/carers refuse to engage with FCAMHS;
* No statutory service is involved in supporting the child;
* No statutory service will agree to hold the child's case open for a minimum of six months.
* Currently involved in another psychological intervention research study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 632 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Reactive and Proactive Aggression Questionnaire (child reported) | Completed at baseline and six months post-baseline (primary endpoint).
  The primary outcome is aggression and violent behaviour measured by the self-reported Reactive and Proactive Aggression Questionnaire. The RPQ combines two subscales, one measuring reactive aggression (12 items), the other proactive aggression (11 items). Each item is scored on a three-point scale from 0 (never) to 2 (often). Item scores from each subscale are added together to produce sub-scale scores (range 0-24 for reactive aggression, and 0-22 for proactive aggression). The total score can range from 0-46.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (child reported) | Completed at baseline and six months post-baseline.
  Five outcomes will be measured using the 30-item Strengths and Difficulties Questionnaire including impact supplement: conduct problems using the conduct problem subscale (5 items); inattention difficulties using the hyperactivity/inattention subscale (5 items); emotional difficulties using the emotional symptoms subscale (5 items); difficulties with peers using the peer relationship problems scale (5 items). Each item is rated on a 3-point scale: Not True = 0, Somewhat True = 1, and Certainly True = 2. For each subscale, scores range from 0 to 10, with higher scores reflecting more difficulties.
  The impact supplement asks participants whether they experience difficulties in emotions, behaviour, concentration, or relationships rated from 'no' to 'severe difficulties'. Further questions ask about interference of these difficulties in areas of life including home, friendships, learning and leisure, rated from 'not at all' to 'a great deal'.
Emotion Awareness Questionnaire (child reported) | Completed at baseline and six months post-baseline.
  Two outcomes will be measured to assess mentalizing using two subscales (10 items) of the Emotion Awareness Questionnaire:
  1. Analyses of emotions (5 items, score 5-15) (sample item: "When I am angry or upset, I try to understand why").
  2. Attending to others' emotions (5 items, score 5-15) (sample item: "It is important to know how my friends are feeling").
  For items in both subscales, responses are scored on a three-point scale from 1 (not true) to 3 (often true).
Systemic Clinical Outcome and Routine Evaluation (SCORE-15) (child reported) | Completed at baseline and six months post-baseline.
  One family outcome will be measured using the total score of the SCORE-15, a 15-item self-report measure designed to assess perceived family functioning across emotional, behavioral, and communication areas. Participants are asked to indicate how well each statement describes their family using a 5-point scale between the range: 1 (Describes us: Very well) to 5 (Describes us: Not at all).
  In addition to the 15-item quantitative scale, the SCORE-15 includes two open-ended, qualitative questions i.e. "What words would best describe your family?" and "What is the problem/challenge that brought you to therapy?".
  Lastly, the SCORE-15 includes three single-item visual analogue scales designed to capture subjective ratings of severity of difficulties (scale of 0 [No problem at all] to 10 [Really bad]), family managing (scale of 0 [very well] to 10 [very badly]), and perceived helpfulness of therapy (scale of 0 [very helpful] to 10 [unhelpful]).
Reactive and Proactive Aggression Questionnaire (parent/carer reported) | Completed at baseline and six months post-baseline.
  One outcome, aggression and violent behaviour, will be measured using a parent/carer version of the RPQ. The RPQ is a 23-item self-report questionnaire designed to assess two subtypes of aggressive behaviour: reactive aggression (12 items) and proactive aggression (11 items). Each item is rated on a 3-point scale indicating frequency of behaviour (0 = Never, 1 = Sometimes, 2 = Often). Subscales range from 0-24 (reactive) and 0-22 (proactive). The total aggression score ranges from 0-46.
Strengths and Difficulties Questionnaire (parent/carer reported) | Completed at baseline and six months post-baseline.
  Five outcomes will be measured using the 30-item parent version of the Strengths and Difficulties Questionnaire including impact supplement: conduct problems using the conduct problem subscale (5 items); inattention difficulties using the hyperactivity/inattention subscale (5 items); emotional difficulties using the emotional symptoms subscale (5 items); difficulties with peers using the peer relationship problems scale (5 items). Each item is rated on a 3-point scale: Not True = 0, Somewhat True = 1, and Certainly True = 2. For each subscale, scores range from 0 to 10, with higher scores reflecting more difficulties.
  The impact supplement asks participants whether their child experiences difficulties in emotions, behaviour, concentration, or relationships rated from 'no' to 'severe difficulties'. Further questions ask about interference of these difficulties in areas of life including home, friendships, learning and leisure, rated from 'not at all' to 'a great deal'.
Systemic Clinical Outcome and Routine Evaluation (SCORE-15) (parent/carer reported) | Completed at baseline and six months post-baseline.
  One family outcome will be measured using the total score of the SCORE-15 as reported by parents/carers. SCORE-15 is a 15-item self-report measure designed to assess perceived family functioning across emotional, behavioural, and communication areas. Participants are asked to indicate how well each statement describes their family using a 5-point scale between the range: 1 (Describes us: Very well) to 5 (Describes us: Not at all).
  In addition to the 15-item quantitative scale, the SCORE-15 includes two open-ended, qualitative questions i.e. "What words would best describe your family?" and "What is the problem/challenge that brought you to therapy?".
  Lastly, the SCORE-15 includes three single-item visual analogue scales designed to capture subjective ratings of severity of difficulties (scale of 0 [No problem at all] to 10 [Really bad]), family managing (scale of 0 [very well] to 10 [very badly]), and perceived helpfulness of therapy (scale of 0 [very helpful] to 10 [unhelpful]).
Health of the Nation Outcome Scales for Children and Adolescents (clinician reported) | Completed at baseline and six months post-baseline.
  Six child outcomes will be measured using six items of the Health of the Nation Outcomes Scales for Children and Adolescents (HoNOSCA) reported by a clinician:
  Disruptive, antisocial or aggressive behaviour; Non accidental self-injury; Substance misuse; Peer relationships; Family life and relationships; School attendance.
  Each item is scored from 0 (no problem) to 4 (severe to very severe problem), with higher scores indicating greater severity. A score of 3 or above on any item indicates a moderate to severe problem.

OTHER OUTCOMES:
Therapeutic alliance (child reported) | Will be assessed at three time points during 6 month reporting period: early therapy (defined as sessions/weeks 1-3), mid-therapy (defined as sessions/weeks 10-13), and late therapy (defined as sessions/weeks 20-24)
  Therapeutic alliance, as a potential mediator or mechanism of change, will be assessed in the intervention arm at three timepoints (early therapy e.g. session 1-3, mid-therapy e.g. session 10-13, and late therapy e.g. session 20-24) using the Session Rating Scale (SRS). The SRS assesses the young person's perceptions of: respect and understanding from the clinician, how much they talk about the topics that matter to them, the clinicians approach or method, and overall acceptability of the session. A visual line is presented with contrasting statements at each e.g. "I did not feel heard, understood and respected", versus "I felt heard, understood and respected", (on the SRS version for 6-12 year olds, the statements are supplemented with a sad face or smiley face, respectively). Participants indicate their experience by placing a mark somewhere along the line. Reponses marked closest to the positive version of the statement (the smiley face) indicate a better therapeutic alliance.
Goal based outcomes (child reported) | Will be assessed at three time points during 6 month reporting period: early therapy (defined as sessions/weeks 1-3), mid-therapy (defined as sessions/weeks 10-13), and late therapy (defined as sessions/weeks 20-24)
  Progress towards goals, as a potential mediator or mechanism of change, will be assessed in the intervention arm at three timepoints (early therapy e.g. session 1-3, mid-therapy e.g. session 10-13, and late therapy e.g. session 20-24) using the goal based outcome (GBO) tool. The GBO enables young people to set up to three goals and rate the extent to which they feel that they have reached their goals on a scale of 0 (no progress) to 10 (fully reached).

CONTACTS AND LOCATIONS:
Locations (11):
- United Kingdom (11):
  - Hampshire and Isle of Wight Healthcare NHS Foundation Trust, Southampton, Calmore
  - South London Community Forensic CAMHS , South London and Maudsley NHS Foundation Trust, Beckenham, Kent
  - Yorkshire and Humber FCAMHS, South West Yorkshire Partnership NHS Foundation Trust, Wakefield, Ouchthorpe Lane
  - South Central Community Forensic CAMHS Team, Oxford Health NHS Foundation Trust, Headington, Oxford
  - South West (North) Community Forensic CAMHS Team, Oxford Health NHS Foundation Trust, Headington, Oxford
  - East Midlands Community Forensic Child & Adolescent Mental Health Service, Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, Porchester Road
  - The North East and North Cumbria Community Forensic Child & Adolescent Mental Health Service, Cumbria, Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle upon Tyne, Upon Tyne and Wear
  - East of England Community FCAMHS Team, Cambridgeshire and Peterborough NHS Foundation Trust, Cambridge
  - Tavistock and Portman NHS Foundation Trust Forensic CAMHS, Tavistock and Portman NHS Foundation Trust, London
  - North West London Forensic Child and Adolescent Mental Health Service , West London NHS Trust, Southall
  - South West FCAMHS, Somerset NHS Foundation Trust, Taunton

IPD SHARING:
Plan to Share IPD: Yes
All anonymous study data (and name, date of birth and postcode) will be securely transferred to the Department for Education (DfE). The DfE will replace all identifying information about the young people who have taken part in the study (their name, date of birth, and postcode) with the young person's unique Pupil Matching Reference number in the DfE's National Pupil Database. The DfE will transfer this data to the YEF archive, which is stored in the Office for National Statistics' Secure Research Service. Access to the anonymised data may be granted to other researchers through controlled procedures governed by the YEF Data Archive.
  Anonymised data will also be retained by the University of Hertfordshire and Anna Freud Centre for up to 10 years to support secondary analysis and related research outputs. This may or may not involve sharing data with other researchers, contributing to a larger data set.

REFERENCES:
- [Background] Hauschild S, Kasper L, Volkert J, Sobanski E, Taubner S. Mentalization-based treatment for adolescents with conduct disorder (MBT-CD): a feasibility study. Eur Child Adolesc Psychiatry. 2023 Dec;32(12):2611-2622. doi: 10.1007/s00787-022-02113-4. Epub 2022 Nov 25. PMID 36434148
- [Background] Taubner S, Hauschild S, Kasper L, Kaess M, Sobanski E, Gablonski TC, Schroder-Pfeifer P, Volkert J. Mentalization-based treatment for adolescents with conduct disorder (MBT-CD): protocol of a feasibility and pilot study. Pilot Feasibility Stud. 2021 Jul 2;7(1):139. doi: 10.1186/s40814-021-00876-2. PMID 34215323
- See also: The MICA study will be hosted on the Anna Freud Research Library platform. — https://www.annafreud.org/research/research-library/
- See also: The Youth Endowment Fund (YEF) archive platform will serve as the hosting platform for anonymised data archived from the MICA study. — https://youthendowmentfund.org.uk/evaluation-data-archive/